CLINICAL TRIAL: NCT05672654
Title: Evaluation of Post-SARS-CoV-2 Vaccinal Response in Immunocompromised Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Responsibility for registering this study lies with the sponsor, DiaSorin, and not with our institution
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: VACCIM
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV Seropositivity; Immunodeficiency; Vaccination Reaction; Covid19
MeSH Terms: conditions — HIV Seropositivity; Immunologic Deficiency Syndromes; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Control group (Active Comparator)
  Interventions: Diagnostic Test: Blood draw
- HIV positive CD4<350 cells/mm^3 (Active Comparator)
  Interventions: Diagnostic Test: Blood draw
- Immune-compromised patients- department rheumatology (Active Comparator)
  Interventions: Diagnostic Test: Blood draw
- Immune-compromised patients- department nephrology (Active Comparator)
  Interventions: Diagnostic Test: Blood draw
- Immune-compromised patients- department neurology (Active Comparator)
  Interventions: Diagnostic Test: Blood draw
- Primary immune deficiency en common variable immunodeficiency (Active Comparator)
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Blood draw

SUMMARY:
The aim of this study is to identify both the humoral immunological response through the detection of induced antibodies and the cellular immunological response through the detection of interferon gamma production by functional CD4+ and CD8+ cells in different groups of immunocompromised patients. For antibody detection, LIAISON® SARS-CoV-2 TrimericS assay (DiaSorin) will be used and for the evaluation of cellular immunity - QuantiFERON SARS-CoV-2 assay (QIAGEN).

DETAILED DESCRIPTION:
The national vaccination campaign against COVID-19 is ongoing and high risk patients are invited. Within the group of high risk patients, there are several groups of people who are for some reason immune-compromised and whose immune system is not functioning adequately. As vaccines against COVID-19 have become available in Europe as a matter of urgency, there are currently insufficient or no data available on the generation of post-vaccinal response in different groups of these immunocompromised patients. The theoretical assumption that the generation of post-vaccinal response in these patients is different from that in immunocompetent individuals is valid, as it has been shown for other vaccines, e.g. against influenza and pneumococcal disease, that the use of immunosuppressive treatments such as asrituximab, methotrexate and rituximab suppress the production of neutralising antibodies. It is known that vaccines against COVID-19 are also capable of inducing a clear functional cellular response in addition to neutralising antibody production, the modalities of which are also insufficiently or not known in these patients.

As mentioned is the goal of VACCIm to identify both the humoral immunological response through the detection of induced antibodies and the cellular immunological response through the detection of interferon gamma production by functional CD4+ and CD8+ cells in different groups of immunocompromised patients.

Within this prospective observational study, serum samples (for subsequent measurement with LIAISON® SARS-CoV-2 TrimericS assay) and lithium-heparin whole blood samples (for subsequent measurement with QuantiFERON SARS-CoV-2 assay) will be collected from control immune-competent individuals and immune-compromised patients within the following groups:

* Common variable immunodeficiency disorders and primary immunodeficiency disorders
* HIV-positive patients with CD4 < 350 cells/mm3
* Immune-compromised patients in rheumatology, neurology and nephrology

In order to assess both humoral and cellular responses as fully as possible, both measurements are performed at the following time points:

T0: before (=prior) or at time of first dose of vaccine T1: 21-28 days after first dose of vaccine T2: at least 10 days after second dose of vaccine T3: after 3 months after second dose of vaccine T4: after 6 months from second dose of vaccine T5: after 12 months from second dose of vaccine

ELIGIBILITY:
Inclusion Criteria:

Following patient groups receiving the Pfizer vaccine

* HIV-positive patients with CD4 < 350 cellen/mm3
* Common variable immunodeficiency disorders en primary immunodeficiency disorders
* Immune-compromised patients hospitalized at rheumatology/neurology/nephrology

Exclusion Criteria:

* patients receiving a different of vaccine

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Humoral immune response | prior or at the time of first dose of vaccine until 12 months after second dose of vaccine
  Detection of Antibodies
Cellular immune response | prior or at the time of first dose of vaccine until 12 months after second dose of vaccine
  DetectionINF-gamma by functional CD4+ and CD8+ cells

CONTACTS AND LOCATIONS:
Locations (1):
- UH Ghent, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided